CLINICAL TRIAL: NCT01621516
Title: Measurement of ß-cell Function and Insulin Sensitivity in Non-diabetic Patients With En-bloc Liver, Pancreas and Small Bowel Transplant Using a Hyperglycemic Clamp
Brief Title: Measurement of the Pancreas Function in Patients With More Than One Pancreas After Liver and Small Bowel Transplantation
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, prof. Pieter Gillard, prof. dr., KU Leuven
Other Study IDs: BCFTX 001
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes; Insulin Resistance; Liver/Small Bowel Transplant
Keywords: Beta-cell function; Liver/small bowel transplant; Donor pancreas; Diabetes; Long-term immunesuppression
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy controls: 10 healthy volunteers
- Solitary small bowel transplant patients: 3
- Liver/small bowel transplant patients: 3

SUMMARY:
Under chronic immunosuppressive and corticosteroid therapy, transplant patients have a tendency to develop in the long-term diabetes. Patients who have received extra pancreatic tissue with their liver and small bowel transplantation have not yet developed insulin resistance or diabetes mellitus. We would like to investigate to which level insulin secretory capacity the extra pancreas together with the native pancreas has in these transplant patients using the hyperglycemic clamp. These data will be compared with the data obtained from healthy controls.

DETAILED DESCRIPTION:
The glycemic control in type 1 diabetic recipients of islet cell grafts is correlated with the ß-cell mass. In the standard technique for liver/small bowel transplant procedure previously described by Grant et al, the pancreas was removed. This surgical method was modified by Sudan et al and the donor pancreas was transplanted intact in these non-diabetic patients. Under chronic immunosuppressive and corticosteroid therapy, these patients with extra ß-cell mass have not developed insulin resistance or diabetes mellitus. To which level insulin secretory capacity the extra pancreas allograft together with the native pancreas has in these transplant patients are not yet known.

Among the measures of pancreatic ß-cell-secretory capacity, the first-phase and steady state insulin secretion from the hyperglycemic clamp studies are believed to give the most robust estimates. Moreover, the hyperglycemic clamp and the euglycemic clamp yield comparable estimates of insulin sensitivity and, so that under appropriate conditions, the hyperglycemic clamp technique may be used to assess both insulin sensitivity and insulin secretion in the same individual in a single experiment.

ELIGIBILITY:
Inclusion Criteria:

* Liver/small bowel transplant patients with partial or whole pancreas
* Solitary small bowel transplant patients
* Insulin independent (no diabetes mellitus)
* Maintenance IS with Tacrolimus/Azathioprine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Liver/small bowel transplant patients with partial or whole pancreas (n = 3):
  Solitary small bowel transplant patients (n=3)
  * Insuline independen (no diabetes mellitus)
  * Maintenance IS with Tacrolimus/Azathioprine
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in the stimulated serum C-peptide leveS (mean area under the curve [AUC] after hypercemic clamp test | One time
  1. Sampling before glucose infusion (-30 to 0 minutes)
  2. Glucose infusion (0 to 14 minutes)
     - increase of glycemia acutely to 180 mg/dL in approx. 14 min.
  3. Clamping at glycemia of 180 mg/dL (15 to 150 minutes)
     * maintain glycemia at 180 mg/dL till 150 min. after start glucose infusion
     * blood sample for measurement of glycemia, proinsulinemia and C-peptide at 120, 135 and 150 minutes (n= 3x5 ml) for evaluation of second-phase insulin release
  4. Intravenous injection of 1 mg glucagon (150 to 170 minutes)